CLINICAL TRIAL: NCT00609115
Title: Sub-Acute Stroke Rehabilitation With Assisted Movement With Enhanced Sensation
Brief Title: Sub-Acute Stroke Rehabilitation With AMES
Acronym: AMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AMES Technology (Industry)
Collaborators: Northwest Medical Rehabilitation, Spokane, WA (Unknown); Emory University (Other); University of California, San Francisco (Other); Shirley Ryan AbilityLab (Other); Eisenhower Medical Center (Other); Legacy Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CT001
Record Dates: First submitted 2007-12-27; First posted 2008-02-06 (Estimated); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-02

CONDITIONS: Cerebrovascular Stroke
Keywords: Sub-acute care; Robotics
MeSH Terms: conditions — Stroke | interventions — Cross-Over Studies

STUDY DESIGN:
Intervention Model Description: Single crossover for only the control group participants from the controlled part of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test-Phase 1 (Experimental): The Test Group receives 18 half-hour AMES (Assisted Movement with Enhanced Sensation) treatments with the AMES device (Test) in which the hand or wrist is moved, and the subject assists the motion while vibration (60 pulses/sec) is applied to the lengthening muscle. Sessions to be scheduled preferably 2 to 3 times per week, with the 18 sessions to be completed within the 6 month anniversary date of the subject's stroke.
  Interventions: Device: AMES device (test)
- Control-Phase 1 (Sham Comparator): Eighteen treatment sessions for each qualifying subject limb using the AMES device (sham) programed to provide placebo therapy. Each treatment session consisting of 30 minutes of sham therapy. Sessions to be scheduled preferably 2 to 3 times per week, with the 18 sessions to be completed within the 6 month anniversary date of the subject's stroke.
  Interventions: Device: AMES device (sham)
- Crossover-Phase 2 (Active Comparator): Original Control Group receives 18 half-hour crossover treatments with the AMES device (Crossover) in which the hand or wrist is moved, and the subject assists the motion while vibration (60 pulses/sec) is applied to the lengthening muscle. Sessions to be scheduled preferably 2 to 3 times per week with each session one-half hour in length.
  Interventions: Device: AMES device (crossover)

INTERVENTIONS:
Device: AMES device (test) — Eighteen treatment sessions for each qualifying subject limb using the AMES device. Each treatment session being 30 minutes long. Sessions to be scheduled preferable 2 to 3 times per week, with the 18 sessions to be completed within the 6 month anniversary date of the subject's stroke.
  Arms: Test-Phase 1
Device: AMES device (sham) — Eighteen treatment sessions for each qualifying subject limb using the AMES device (sham) in which the limb is moved, but no active assistance is provided by the subject and the vibration is delivered at a very low frequency to the shortening (i.e., rather than lengthening) muscle. Each treatment session to provide thirty minutes of the placebo form of AMES therapy.
  Arms: Control-Phase 1
Device: AMES device (crossover) — Eighteen treatment sessions for each qualifying subject limb using the AMES device. Each treatment session being 30 minutes long. Sessions to be scheduled preferable 2 to 3 times per week, with the 18 sessions to be completed as soon as possible after the completion of Arm C-1 Sham Comparator.
  Arms: Crossover-Phase 2

SUMMARY:
The AMES device is designed to produce functional cortical changes by:(1) assisting the subject as he/she attempts to move the limb (assisted movement) and (2) enhancing movement sensation by vibrating the muscles during movement (enhanced sensation). The primary hypothesis is that the combination of assisted movement and enhanced sensation from muscle vibration can increase the amount of motor recovery in individuals disabled by a stroke.

DETAILED DESCRIPTION:
Approximately 700,000 U.S. citizens have a stroke each year with about half ending up with significant motor disabilities. There are an estimated 5 million stroke survivors in the U.S., making strokes the leading cause of long-term disability in the U.S.. Existing rehabilitation therapies have not been effective in returning all stroke survivors to full motor recovery.

The AMES device was designed to be able to provide therapy for the hand (fingers/wrist). In this 18 treatment sessions, double-blinded, control study, AMES therapy will be provided in addition to the usual physician-ordered rehabilitation during the sub-acute period following a stroke. Those control subject who complete the Phase 1 placebo sessions will have the opportunity to cross-over to participate in a AMES treatment group for a Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Hemispheric stroke (ischemic or hemorrhagic), cortical or sub-cortical, documented by either a CT or MRI scan and associated with residual weakness in the arm and/or leg.
* First time ever stroke or previous stroke with complete resolution of motor deficit, occurring ≤4 months prior to subject enrollment.
* Age 18-80 years old.
* Moderate to severe lower-extremity paresis (defined as a leg motor Fugl-Meyer score of ≥6 and ≤22 out of a possible 34.
* Moderate to severe upper-extremity paresis (defined as an arm motor Fugl-Meyer score of ≥6 and ≤43 out of a possible 66.
* Visible voluntary movement of the ankle in at least one direction: dorsiflexion or plantarflexion for the ankle and flexion or extension for the hand.
* At least partially functioning proprioception from the paretic arm or leg-capable of correctly identifying, ≥70% of the time, the direction of passive joint rotation (i.e., flexion-extension) with eyes closed.
* Physically and cognitively capable of consenting to and complying with the protocol.
* Score of <19 out of 63 on the 21-question version of the Beck Depression Inventory.
* Subject or legally authorized representative must be capable of providing informed consent.-

Exclusion Criteria:

* Complete flaccidity of the hand, wrist, and ankle.
* Pathological neurological/physical conditions, other than stroke, impairing the function of the impaired arm or leg or resulting in pain in either the arm or leg.
* Spinal cord injury, arthritis, or fractures of affected limbs that have resulted in loss of range of motion.
* Peripheral nerve injury or neuropathy resulting in significant motor or sensory loss in the limb being considered for testing.
* Cardiopulmonary compromise including but not limited to uncontrolled hypertension or angina, deep vein thrombosis, decompensated congestive heart failure, myocardial infarction, heart irregularities, or exercise intolerance.
* Major active psychiatric disorder.
* Severe apraxia; inability to understand verbal (English) directions; or inability to communicate adequately with study personnel.
* Size of arm or leg incompatible with the AMES device.
* Severe contractures or decreased range of motion that would prohibit comfortable positioning or tolerance of the device
* Skin condition not able to tolerate use of the AMES device.
* Any progressive neurodegenerative disorder affecting the motor system.
* Uncontrolled seizure disorder.
* Current abuse of alcohol or drugs.
* Terminal illness with anticipated survival of <12 months.
* Current or planned concurrent participation in another study or clinical trial.
* NIH Stroke Scale, following scores: Item 1a > 0; Item 1c > 0; Item 2 > 0; Item 3 > 0; Item 9 > 2; Item 10 > 1; Item 11 > 1 (based on exam by Study Physician).
* Intent to receive Botox injections, initiation of antispasmodic medication, or use any other robotic (e.g., MANUS, Locomat) or stimulation device (e.g., Bioness) while participating in the AMES trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Cordo, PhD, Study Director — AMES Technology Inc./ Oregon Health and Science University
Locations (5):
- United States (5):
  - Eisenhower Medical Center, Rancho Mirage, California
  - UCSF School of Medicine- Physical Therapy and Rehabilitation, San Francisco, California
  - Emory University Dept of Rehabilitation Medicine/School of Medicine, Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - NW Medical Rehabilitation, Spokane, Washington

REFERENCES:
- [Derived] Cordo P, Wolf S, Rymer WZ, Byl N, Stanek K, Hayes JR. Assisted Movement With Proprioceptive Stimulation Augments Recovery From Moderate-To-Severe Upper Limb Impairment During Subacute Stroke Period: A Randomized Clinical Trial. Neurorehabil Neural Repair. 2022 Mar;36(3):239-250. doi: 10.1177/15459683211063159. Epub 2022 Jan 24. PMID 35067125
- See also: Study sponsor AMES Technology, Inc. website — http://amesdevices.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants enrolled and assigned to the test or control group dropped out of the study. Each drop-out was encouraged to participate in a post-treatment evaluation, even though the standard course of treatment (i.e., 18 one-half hour sessions) was not completed. The data from participants who complied with this request were included in the analysis. Those not complying were not included. However, baseline values reported here include baseline data from all drop-out participants.
Period: Controlled Period
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Started | 44 | 39 | 0
Completed | 38 | 35 | 0
Not Completed | 6 | 4 | 0
Period: Crossover Period
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Started | 0 | 0 | 27
Completed | 0 | 0 | 22
Not Completed | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test-Phase 1 | Control-Phase 1 | Total
Number analyzed (Participants) | 44 | 39 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.7) | 57.7 (12.9) | 57.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 29 | 23 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 36 | 32 | 68
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 11 | 23
  White | 25 | 22 | 47
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 3 | 7
Stroke Type [Count of Participants; unit: Participants]
  Ischemic | 37 | 34 | 71
  Hemorrhagic or Ischemic Plus Hemorrhagic | 7 | 5 | 12
Study Site [Count of Participants; unit: Participants]
  Site 1 | 8 | 7 | 15
  Site 2 | 1 | 0 | 1
  Site 3 | 10 | 9 | 19
  Site 4 | 0 | 1 | 1
  Site 5 | 5 | 3 | 8
  Site 6 | 20 | 19 | 39
Time Since Stroke at Baseline [Mean (Standard Deviation); unit: Weeks] | 11.8 (5.7) | 11.3 (5.0) | 11.5 (5.4)
Active Motion Test Grasp [Mean (Standard Deviation); unit: Seconds] — Performance analysis was based on the total time (in seconds) during the test that the subject was able to keep the tracking line, which represented the subject's joint angle, within the moving target. Intent is to report a change from baseline. Population: Two drop-out participants did not attend the first 3 training sessions and, therefore, did not contribute baselines scores on this test.
  Seconds
    number analyzed (Participants) | 44 | 37 | 81
    (all) | 9.8 (4.9) | 10.0 (6.7) | 9.9 (5.5)
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — This baseline measure was obtained during each candidate subject's evaluation of eligibility for enrollment in the study. Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Scores were obtained for each of 7 categories of evaluation and summed for a final score. The range of possible scores for this measure is 0-66, with 0 representing no motor function and 66 representing normal motor function.
  units on a scale | 20.9 (9.9) | 23.7 (11.2) | 22.5 (10.9)
Spasticity (Modified Ashworth) Scale [Mean (Standard Deviation); unit: units on a scale] — Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Spasticity is represented by the sum of 4 individual measures (finger and wrist flexion, finger and wrist extension, elbow flexion, and elbow extension). Each individual measure represents the resistance of the joint to passive motion. The range of possible scores for each joint is 0-5 with 5 representing the most resistance and 0 representing normal resistance.
  units on a scale | 4.1 (3.0) | 4.6 (3.0) | 4.3 (3.0)
Strength Grasp Flexion [Mean (Standard Deviation); unit: Newton meters] — Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Maximum grasping strength was measured 3 times (trials), in succession, at the end of each training session. The baseline measure of grasp flexion strength consists of the average of the 9 "squeeze" strength trials performed during the first 3 training sessions (i.e., 3 trials in each). Population: Two control group drop-out participants did not contribute baselines scores on this test.
  Newton meters
    number analyzed (Participants) | 44 | 37 | 81
    (all) | 14.6 (14.3) | 16.4 (19.9) | 15.4 (16.8)
Strength Wrist Flexion [Mean (Standard Deviation); unit: Newton-meters] — Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Maximum wrist flexion strength was measured 3 times (trials), in succession, at the end of each training session. The baseline measure of wrist flexion strength consists of the average of the 9 wrist flexion strength trials performed during the first 3 training sessions (i.e., 3 trials in each). Population: Two test group drop-out and one control group drop-out participants did not contribute baselines scores on this test.
  Newton-meters
    number analyzed (Participants) | 42 | 38 | 80
    (all) | 31.7 (27.4) | 36.5 (39.4) | 33.9 (33.0)
Strength Grasp Extension [Mean (Standard Deviation); unit: Newton-meters] — Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Maximum hand-opening strength was measured 3 times (trials), in succession, at the end of each training session. The baseline measure of finger-thumb extension strength consists of the average of the 9 "hand-opening" strength trials performed during the first 3 training sessions (i.e., 3 trials in each). Population: Two control group drop-out participants did not attend the first 3 training sessions and, therefore, did not contribute baselines scores on this test.
  Newton-meters
    number analyzed (Participants) | 44 | 37 | 81
    (all) | 2.6 (4.6) | 2.5 (6.2) | 2.6 (5.3)
Strength Wrist Extension [Mean (Standard Deviation); unit: Newton-meters] — Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Maximum wrist extension strength was measured 3 times (trials), in succession, at the end of each training session. The baseline measure of grasp flexion strength consists of the average of the 9 wrist extension strength trials performed during the first 3 training sessions (i.e., 3 trials in each). Population: One test group drop-out and two control group drop-out participants did not contribute baselines scores on this test.
  Newton-meters
    number analyzed (Participants) | 43 | 37 | 80
    (all) | 11.3 (14.8) | 10.5 (14.6) | 10.9 (14.7)
Stroke Impact Scale [Mean (Standard Deviation); unit: units on a scale] — A self-reporting assessment of functionality across 8 different domains (e.g., strength, communication, memory). Each domain consists of 4-10 questions,each question scored from 1-5 representing the spectrum from "could not do it at all" to "not difficult at all." A total score for all 8 domains is obtained as follows: Total=[(raw score-lowest possible score)/possible raw score] x 100. Intent is to report a change from baseline. Population: A site inadvertently omitted this test with one test group subject and one control group subject.
  units on a scale
    number analyzed (Participants) | 43 | 38 | 81
    (all) | 506.8 (80.9) | 500.3 (92.9) | 503.8 (86.5)
Rancho Los Amigos Functional Test [Mean (Standard Deviation); unit: Number of tasks completed] — This test measures the ability to manipulate objects in everyday functional tasks. A total of 17 different tasks are attempted by each subject. The test quantifies both the ability to perform the task at all and, if performed, the quality of performance. Only the number of tasks that could be performed at any level were analyzed. The criteria distinguishing non-performance from performance are well defined. Intent is to report change from baseline. Population: A site inadvertently omitted this test on one control group participant.
  Number of tasks completed
    number analyzed (Participants) | 44 | 38 | 82
    (all) | 4.8 (3.7) | 5.9 (4.5) | 5.3 (4.1)
Active Motion Wrist Test [Mean (Standard Deviation); unit: Seconds] — Performance analysis was based on the total time (in seconds) during the test that the subject was able to keep the tracking line, which represented the subject's joint angle, within the moving target. Intent is to report change from baseline. Population: One test group drop-out and two control group drop-out participants did not attend the first 3 training sessions and, therefore, did not contribute baselines scores on this test.
  Seconds
    number analyzed (Participants) | 43 | 37 | 80
    (all) | 17.6 (10.7) | 17.3 (11.3) | 17.4 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment Upper Limb Portion
Description: Comprehensive measure of upper limb impairment; minimum score = 0, maximum score = 66; higher score means better outcome. Outcome measure represents the difference between post-treatment and baseline (i.e., change score). Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: Post-treatment-Phase 1 (month 3-6 post-stroke), post-crossover treatment-Phase 2 (month 5-7 post-stroke).
Population: Participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
units on a scale | 10.8 (7.4) | 6.4 (7.7) | 4.7 (6.7)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.010, ANCOVA; Effect size = 0.65
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.003, ANCOVA; Effect = 0.71

2. Secondary Outcome: Stroke Impact Scale
Description: Activities of daily living questionnaire for stroke patients. Minimum overall score = 0, maximum overall score = 800. Higher scores mean better outcome. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: Post-treatment-Phase 1 (month 3-6 post-stroke), post-crossover treatment-Phase 2 (month 5-7 post-stroke).
Population: Participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
units on a scale | 14.6 (28.5) | 10.7 (15.2) | 46.2 (32.4)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 1.00, ANCOVA — The reported p-value was calculated; Effect Size = 0.00
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.06, ANCOVA; Effect Size = -0.29

3. Secondary Outcome: Rancho Los Amigos Functional Test
Description: Upper limb functional movement. Outcome measure indicates how many of 17 functional tasks could be completed. Minimum score = 0, maximum score = 17. Higher number means better outcome. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: Post-treatment-Phase 1 (month 3-6 post-stroke), post-crossover treatment-Phase 2 (month 5-7 post-stroke).
Population: participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
units on a scale | 3.5 (4.3) | 2.1 (3.4) | -0.6 (2.0)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.17, ANCOVA; Effect Size = 0.33
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.17, ANCOVA; Effect Size = 0.40

4. Secondary Outcome: Spasticity (Modified Ashworth) Scale
Description: Joint impedance of the fingers+wrist combined and that of the elbow. Outcome measure consists of the sum of 4 scores: (1) hand/wrist flexion, (2) hand/wrist extension, (3) elbow flexion, (4) elbow extension. Minimum value = 0, maximum value = 20. Higher score means worse outcome. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: Post-treatment-Phase 1 (month 3-6 post-stroke), post-crossover treatment-Phase 2 (month 5-7 post-stroke).
Population: participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
units on a scale | 0.0 (2.1) | -0.6 (2.9) | -0.6 (2.0)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.83, ANCOVA; Effect Size = 0.05
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.83, ANCOVA; Effect Size = -0.27

5. Secondary Outcome: Active Motion Test Grasp
Description: Ability to track a moving target with active grasp extension and flexion, measured as the total time in the target, in seconds. Outcome measure represents the change score from baseline to post-treatment. Minimum score = 0, maximum score = 40 s. Higher scores indicate better outcome. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: Prior to each treatment session. Post-treatment-Phase 1 (month 3-6 post-stroke), post-crossover treatment-Phase 2 (month 5-7 post-stroke).
Population: participants
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
seconds | 2.6 (4.1) | 1.5 (4.4) | 2.4 (6.3)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.28, ANCOVA; Effect Size = 0.25
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.09, ANCOVA; Effect Size = 0.38

6. Secondary Outcome: Active Motion Wrist
Description: Ability to track a moving target with active wrist extension and flexion, measured as the total time in the target, in seconds. Outcome measure represents the change score from baseline to post-treatment. Minimum score = 0, maximum score = 40 s. Higher scores indicate better outcome. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: as for outcome 5
Population: participants
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
seconds | 4.4 (5.8) | 2.7 (4.4) | 1.9 (5.2)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.18, ANCOVA; Effect Size = 0.23
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.10, ANCOVA; Effect Size = 0.37

7. Secondary Outcome: Strength Grasp Flexion
Description: Isometric grasp flexion strength. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: as for outcome 5
Population: participants
Measure: Mean (Standard Deviation); unit: Newton-meter
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
Newton-meter | 26.3 (1.6) | 24.6 (1.7) | 8.5 (11.9)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.45, ANCOVA; Effect Size = 0.18
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.003, ANCOVA; Effect Size = 0.71

8. Secondary Outcome: Strength Grasp Extension
Description: Isometric grasp extension strength. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: as for outcome 5
Population: participants
Measure: Mean (Standard Deviation); unit: Newton-meter
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
Newton-meter | 4.2 (0.6) | 4.9 (0.6) | 4.3 (7.6)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.47, ANCOVA; Effect Size = -0.17
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.015, ANCOVA; Effect Size = 0.77

9. Secondary Outcome: Strength Wrist Flexion
Description: Isometric wrist flexion strength. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: as for outcome 5
Population: participant
Measure: Mean (Standard Deviation); unit: Newton-meter
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
Newton-meter | 53.8 (2.6) | 46.2 (2.7) | 16.2 (21.1)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.05, ANCOVA; Effect Size = 0.48
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.002, ANCOVA; Effect Size = 0.56

10. Secondary Outcome: Strength Wrist Extension
Description: Isometric wrist extension strength. Intent is to report a change from baseline to post-treatment Phase 1 for both Test Group subjects and Control Group subjects, and to report a change from post-treatment Phase 1 to post-crossover treatment Phase 2 for Control Group subjects who elected to cross over.
Time Frame: as for outcome 5
Population: participant
Measure: Mean (Standard Deviation); unit: Newton-meter
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
Number analyzed (Participants) | 38 | 35 | 22
Newton-meter | 20.7 (1.5) | 18.3 (1.6) | 8.9 (19.8)
Statistical Analysis 1: Comparison: Test-Phase 1 vs Control-Phase 1; Test type: Superiority; p = 0.27, ANCOVA; Effect Size = 0.26
Statistical Analysis 2: Comparison: Control-Phase 1 vs Crossover-Phase 2; Test type: Superiority; p = 0.045, ANCOVA; Effect Size = 0.45

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of each participant's period of participation in the study. For participants in the Test group, and those in the Control group who chose not to cross over, the time frame was 6-9 weeks. For those Control group participants who crossed over, the time frame was 9-14 weeks.
Arm/Group | Test-Phase 1 | Control-Phase 1 | Crossover-Phase 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/39 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/39 | 0/27
Other Adverse Events (participants affected / at risk) | 1/44 | 2/39 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test-Phase 1 (N=44) | Control-Phase 1 (N=39) | Crossover-Phase 2 (N=27)
Skin abrasion from vibrator probe (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No